CLINICAL TRIAL: NCT06009965
Title: Establishment of an Efficacy and Relapse Prediction System for Immunosuppressants Combined With Thrombopoietin Receptor Agonists in the Treatment of Aplastic Anemia
Brief Title: Efficacy of IST Combined With TPO-RA in the Treatment of AA and Establishment of a Recurrence Prediction System
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-01
Record Dates: First submitted 2023-08-06; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Aplastic Anemia; CSA; Drug Therapy
Keywords: Aplastic Anemia; CsA; ATG; TPO-RA
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe aplastic anemia group (Experimental): CsA: 3-5 mg/kg/day, monitor trough concentration monthly, maintain trough concentration at 100-200 ng/ml.ATG: rabbit anti-thymocyte immunoglobulin (r-ATG) 3 mg/kg/d x 5 days or porcine anti-lymphocyte immunoglobulin ((p-ATG) 25 mg/kg/d x 5 days.TPO-RA: Heptapepto-Papa 7.5 mg qd to start. Monitor blood every 2 weeks and if ineffective, increase by 1 tablet every 2 weeks up to a maximum of 6 tablets (15mg) qd.
  Interventions: Drug: CsA+ATG+Herombopag
- Non-severe aplastic anemia group (Experimental): CsA: 3-5 mg/kg/day, monitor trough concentrations monthly, maintain trough concentrations at 100-200 ng/ml.TPO-RA: Start with Hetropoxyphene 7.5 mg qd, monitor blood every 2 weeks, and if ineffective, increase by 1 tablet every 2 weeks up to a maximum of 6 tablets (15 mg) qd.
  Interventions: Drug: CsA+Herombopag

INTERVENTIONS:
Drug: CsA+ATG+Herombopag — CsA: 3-5 mg/kg/day, monitor trough concentration monthly, maintain trough concentration at 100-200 ng/ml.ATG: rabbit anti-thymocyte immunoglobulin (r-ATG) 3 mg/kg/d x 5 days or porcine anti-lymphocyte immunoglobulin ((p-ATG) 25 mg/kg/d x 5 days.TPO-RA: Heptapepto-Papa 7.5 mg qd to start. Monitor blood every 2 weeks and if ineffective, increase by 1 tablet every 2 weeks up to a maximum of 6 tablets (15mg) qd.
  Other Names: SAA group intervention treatment
  Arms: Severe aplastic anemia group
Drug: CsA+Herombopag — CsA: 3-5 mg/kg/day, monitor trough concentrations monthly, maintain trough concentrations at 100-200 ng/ml.TPO-RA: Start with Hetropoxyphene 7.5 mg qd, monitor blood every 2 weeks, and if ineffective, increase by 1 tablet every 2 weeks up to a maximum of 6 tablets (15 mg) qd.
  Other Names: NSAA group intervention treatment
  Arms: Non-severe aplastic anemia group

SUMMARY:
In this study, investigators intend to prospectively study treatment-naive AA patients (including SAA and NSAA) who are non-transplant candidates in northern China. Patients with SAA receive ATG+CsA+Herombopag, and patients with NSAA receive CsA+ Herombopag. Investigators explored possible indicators of participants' predictive efficacy and built predictive models. After the participants achieved response, they used a tapering regimen, observed relapse and clonal evolution, and developed a predictive model of relapse.

DETAILED DESCRIPTION:
1) Patients in the SAA group: CsA: 3-5mg/kg/day, monitor the trough concentration every month, and maintain the trough concentration at 100-200ng/ml. ATG: rabbit anti-thymocyte immunoglobulin (r-ATG) 3mg/kg/d×5 days, or porcine anti-lymphocyte immunoglobulin ((p-ATG) 25mg/kg/d×5 days; TPO-RA: Herombopag starts at 7.5 mg qd, monitor the blood picture every 2 weeks, if the effect is not good, add 1 tablet every 2 weeks, up to 6 tablets (15 mg) qd.

Patients in the NSAA group: CsA: 3-5mg/kg/day, monitor the trough concentration every month, and maintain the trough concentration at 100-200ng/ml. TPO-RA: start with 7.5mg qd of Herombopag, monitor the blood picture every 2 weeks, if the effect is not good, add 1 tablet every 2 weeks, up to 6 tablets (15mg) qd.

(2) Those who are effective after 6 months of treatment continue to receive sufficient CsA treatment for at least 1.5 years, and then slowly reduce the dose until the end of the reduction. Those who fail to withdraw from the clinical trial.

(3) Participants who achieve CR or PR after treatment, but when the curative effect does not increase after 3 months of maintenance treatment, start to reduce the dose of Herombopag, and reduce one tablet every 3 months until the reduction stops. If recurrence occurs, recover Up to the last dose or even increase the dose, after reaching the best curative effect, reduce one tablet every 3 months until the reduction stops, and those who cannot recover are defined as relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, gender is not limited
2. Definite diagnosis of AA
3. No HSCT indication or unconditional HSCT
4. SAA/VSAA patients were willing to accept ATG+CsA+TPO-RA treatment, NSAA was willing to accept CsA+TPO-RA treatment, and were willing to follow up regularly
5. Baseline serum transaminase, total bilirubin and serum creatinine were less than 1.5 times the normal value
6. Baseline liver and kidney function was less than 1.5 times the normal value
7. Eastern Cancer Cooperation Group (ECOG) score status 0-2
8. Agree to sign the consent form

Exclusion Criteria:

1. Congenital AA
2. Cytogenetic evidence of clonal hematologic bone marrow disease
3. PNH clone ≥50%
4. Allergic to ATG, cyclosporine and hexapopal in the past
5. Uncontrolled infection or bleeding at enrollment
6. Received hematopoietic stem cell transplantation (HSCT) before enrollment
7. Any concomitant malignancy within 5 years, except for local skin basal cell carcinoma
8. A history of thromboembolic events, myocardial infarction, or stroke (including antiphospholipid antibody syndrome); Currently using anticoagulants
9. Pregnant or lactating women
10. Situations considered unsuitable for clinical research by other researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 24 weeks after treatment
  Overall response rate
24-month recurrence rate | 96 weeks after treatment
  .24-month recurrence rate

SECONDARY OUTCOMES:
Overall response rate | 56 weeks after treatment
  Overall response rate
36-month recurrence rate | 144 weeks after treatment
  36-month recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Bing Bing, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: email request